CLINICAL TRIAL: NCT01545401
Title: Empowering Primary Care Providers and Patients to Improve Chronic Disease Outcomes: The EMPOWER Participatory Action Research (EMPOWER - PAR)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Collaborators: Ministry of Education, Malaysia (Other Government); Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Sharmila MKL, Dr, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMRR-11-250-8769
Record Dates: First submitted 2012-03-01; First posted 2012-03-06 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes Mellitus; Hypertension (Without Type 2 Diabetes Mellitus)
Keywords: chronic disease management; Chronic Care Model; multifaceted intervention; primary care; type 2 diabetes mellitus; hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EMPOWER-PAR Intervention (Experimental): The intervention arm receives the EMPOWER-PAR intervention package consisting of:
  1. Chronic Disease Management (CDM) Training Workshops for the staff in the respective clinics
  2. The Global CV Risks Self-Management Booklet (patient self-management tool) to empower patients to self-manage their CV risk factors
  3. Facilitation and support of the staff in these clinics so that they may implement the interventions
  Interventions: Other: EMPOWER-PAR Intervention
- Control (No Intervention): The control arm continues with usual care.
  The EMPOWER-PAR intervention package will be made available after the trial ends.

INTERVENTIONS:
Other: EMPOWER-PAR Intervention — Implementation process is conducted in 3 phases:
  I. Phase 1: Formation and training of the CDM team
  II. Phase 2: Distributions of the intervention tools
  * Global CV Risks Self-Management Booklets
  * CPG to aid clinical decision making
  III. Phase 3: Facilitation and support to implement the intervention
  Arms: EMPOWER-PAR Intervention

SUMMARY:
BACKGROUND

Chronic disease management (CDM) presents enormous challenges to the primary care workforce due to the rising epidemic of cardiovascular risk factors. The Chronic Care Model (CCM) was proven effective in improving chronic disease outcomes in developed countries. Evidence that this model works in developing countries is still scarce. Therefore, the aim of this study is to evaluate the effectiveness of the EMPOWER-PAR intervention (multifaceted CDM strategies based on the CCM) in managing type 2 diabetes mellitus (T2DM) and hypertension (HPT), using readily available resources in the Malaysian public primary care setting.

METHODS

This is a pragmatic cluster randomised controlled trial - participatory action research which is currently being conducted in 10 public primary care clinics in Selangor and Kuala Lumpur, Malaysia. Five clinics are randomly selected to provide the EMPOWER-PAR intervention for 1 year, while the other 5 clinics continued with usual care. Each clinic recruits consecutive T2DM and HPT patients who fulfil the inclusion and exclusion criteria over a 2-week period.

The EMPOWER-PAR intervention consists of creating/strengthening a multidisciplinary CDM Team; and training the team to utilise the Global CV Risks Self-Management Booklet to support patient care and reinforcing them to utilise relevant clinical practice guidelines to aid management and prescribing.

For T2DM, primary outcome is the change in the proportion of patients achieving target HbA1c of <6.5%. For HPT without T2DM, primary outcome is the change in the proportion of patients achieving target blood pressure of <140/90 mmHg. Secondary outcomes include the proportion of patients achieving targets serum lipid profile, body mass index and waist circumference. Other outcome measures include medication adherence levels, process of care and prescribing patterns. Patients' assessment of their chronic disease care, providers' perception, attitude and perceived barriers in delivering the care and cost-effectiveness of the intervention are also evaluated.

CONCLUSION

Results from this study will provide objective evidence of the effectiveness and cost-effectiveness of a multifaceted intervention based on the CCM in resource constraint public primary care setting. It is hoped that the evidence will instigate the much needed primary care system change in Malaysia.

DETAILED DESCRIPTION:
HYPOTHESES

The primary hypothesis for T2DM patients is that the proportion achieving target HbA1c of <6.5% would improve with the EMPOWER-PAR intervention. The primary hypothesis for HPT patients without T2DM is that the proportion achieving target BP of <140/90 mmHg would improve with the EMPOWER-PAR intervention.

The secondary hypothesis for T2DM patients is that the proportion achieving target blood pressure (BP) of <130/80 mmHg would improve with the EMPOWER-PAR intervention. The secondary hypotheses for both groups of patients (T2DM and HPT without T2DM) are that the proportions achieving target fasting serum lipid, body mass index (BMI) and waist circumference (WC) would improve with the intervention. Medication adherence levels and patients' perceptions of their experience in receiving chronic disease care are also expected to improve with the intervention. Secondary hypotheses are also made at the primary care providers' level in terms of the process of care and prescribing pattern which are expected to improve with the intervention. Cost-effectiveness analysis and primary care providers' perception, attitude, experience and perceived barriers in implementing the intervention are also explored.

METHODS

* Pragmatic cluster-randomised parallel controlled trial -participatory action research conducted in 10 public primary care clinics from two states in Malaysia which are Wilayah Persekutuan Kuala Lumpur (WPKL) and Selangor (SEL).
* The overall duration of the study is 2 years while the duration of intervention is 1 year.
* Blinding is not possible due to the nature and complexity of the intervention.

Site Recruitment

Site eligibility

All 34 clinics led by Family Medicine Specialists (FMS) in SEL and WPKL are invited to participate in the study and are given the site feasibility assessment form.

To be eligible, the clinics must satisfy all of the following criteria:

i. have a minimum of 500 T2DM patients and 500 HPT patients in the registry. ii. have an FMS who is keen to participate in the study and is willing to lead the implementation of the intervention components in the clinic.

iii. Have the minimum capacity to implement the obligatory components of the EMPOWER-PAR intervention.

iv. located within 70 km from the central laboratory as the blood samples are transported back to the centre for analysis.

Site selection

Site feasibility assessment is conducted to identify eligible clinics. Out of the 34 sites, only 20 fulfil the eligibility criteria to enter the study. These 20 clinics are then matched into 10 pairs according to their geographical locations, staffing and workload. Geographical location is divided into urban and sub-urban areas. Urban area is defined as an area located within a major city, while sub-urban area is defined as an area located surrounding and within commuting distance to a major city. Staffing is defined as the number of doctors and allied health personnel (FMS, medical officers, assistant medical officers, staff nurses, dieticians/nutritionists and pharmacists) working in the clinic. Workload is defined as the average number of patients being seen in the clinic per day.

Multistage randomisation is performed using computer generated tables. The first stage is to randomly select 5 out of the 10 pairs to be included into the study. The second stage is to randomly allocate the clinics into intervention and control arms.

Patient Recruitment

This study recruits consecutive T2DM and/or HPT patients who attend the selected clinic within the 2-week recruitment period. They are given the patient information sheet in the waiting area. Informed consents are obtained from those who are willing to participate. Screening is conducted to identify eligible participants based on the inclusion and exclusion criteria. Eligible patients are then enrolled into the study.

Inclusion criteria

Males and females aged ≥ 18 years who are diagnosed with:

1. T2DM or HPT or both
2. Seen at least once in the last one year at the primary care clinic for the above conditions

Exclusion criteria

1. Type 1 Diabetes Mellitus
2. Receiving renal dialysis
3. Presenting with severe HPT (Systolic BP >180mmHg and/or Diastolic BP >110 mmHg)
4. Diagnosed with conditions resulting in secondary hypertension
5. Diagnosed to have circulatory disorders needing referral to secondary care over the last 1 year e.g. unstable angina, heart attack, stroke, transient ischaemic attacks
6. Receiving shared care between primary and secondary care for complications of T2DM and/or HPT
7. Pregnancy
8. Enrolled in another study

All patients in the intervention arm are required to be seen at least twice by the CDM team of each clinic during the 1-year intervention period. Those who do not comply are considered as lost to follow-up. There is no limit to the number of clinic visits a patient is allowed to make in either arm during the course of the study.

The EMPOWER-PAR INTERVENTION

The study intervention, referred to as the EMPOWER-PAR Intervention, is developed in accordance with the Medical Research Council (MRC) guidance on developing and evaluating complex interventions to improve health outcomes and is implemented at the primary care clinics for a period of 1-year.

The underlying framework in developing the complex intervention for EMPOWER-PAR is based on 6 interrelated elements of the CCM. The 6 elements are 1) organisation of health care (i.e. providing leadership and minimising barriers to care), 2) self-management support (i.e. facilitating skills-based learning and patient empowerment), 3) decision support (i.e. providing guidance for implementing evidence-based care), 4) delivery system design (i.e. coordinating care processes), 5) clinical information systems (i.e. tracking progress through reporting outcomes to patients and providers), and 6) community resources and policies (i.e. sustaining care by using community-based resources).

Three obligatory components which define the EMPOWER-PAR intervention are developed based on 4 interrelated elements of CCM (organisation of health care, delivery system design, self-management support and decision support). These intervention components utilise readily available and existing resources in the Malaysian public primary care setting.

I. Creating/Strengthening a CDM Team-a multidisciplinary team lead by FMS to improve coordination of care for T2DM and/or HPT and co-existing CV risk factors

II. Utilising the Global CV Risks Self-Management Booklet to support patients self-management

III. Utilising the Clinical Practice Guidelines (CPG) for T2DM and HPT to aid management and prescribing

Two optional components of the EMPOWER-PAR intervention are developed based on the other 2 CCM elements (clinical information system and community resources):

I. Utilising clinical information system and conducting clinical audits to track progress through reporting outcomes to patients and providers

II. Utilising community resources to support and sustain care

SAMPLE SIZE CALCULATIONS

The sample size calculation was conducted based on the randomised clustered trial design using PASS software (Copyright (c) 2009 by Dr Jerry L. Hintze, All Rights Reserved).

Sample size calculation for T2DM patients

A sample size of 626 (313 in each arm) is obtained by sampling 10 clusters (5 intervention vs 5 control) with 63 subjects from each cluster to achieve 91% power to detect 25% difference in the proportion of subjects achieving target HbA1c <6.5% from baseline and between the intervention and control groups. The test statistic used is the two-sided Z test (unpooled). The significance level of the test is 0.05. Therefore, after allowing for 25% dropout rate, this study aims to recruit a total sample of 836 T2DM patients at baseline i.e. 418 in each arm and 84 from each clinic.

Sample size calculation for HPT patients without T2DM

A sample size of 438 (219 in each arm) is obtained by sampling 10 clusters (5 intervention vs 5 control) with 44 subjects from each cluster to achieve 88% power to detect 25% difference in the proportion of subjects achieving target BP <140/90 mmHg from baseline and between the intervention and control groups. The test statistic used is the two-sided Z test (unpooled). The significance level of the test is 0.05. Therefore, after allowing for 25% dropout rate, this study aims to recruit a total sample of 584 HPT patients at baseline i.e. 292 in each arm and 58 from each clinic.

STATISTICAL ANALYSIS

The statistical analysis plan to test the primary hypotheses of the study is described. Continuous variables will be described by summary statistics (means and standard deviations) for normally distributed variables. If the distribution is not normal, median with inter-quartile range will be reported instead. Other descriptive statistics, such as minimum and maximum values will be reported when necessary. Categorical (nominal/ordinal) variables will be described by frequencies with percentages. All outcomes are treated as categorical variables (e.g. proportions of patients achieving targets for HbA1c and BP). To assess the differences in the proportions of patients who are able to reach the treatment goals by their intervention strategy, a generalized estimation equation model that adjusts for clustering effects will be used. The model will be an independent working model. Treatment effects will be obtained using the estimated marginal means and differences will be tested using the Wald chi-square tests. The power of the study will be recalculated based on the effect size and after taking into account the clustering effect of the study design. An intention-to-treat analysis will be conducted, and P-values of less than 0.05 will be considered significant. All analyses will be carried out using SPSS (IBM Corp. Released 2011 IBM SPSS Statistics for Windows, Version 20.0. Armonk, NY: IBM Corp.).

ETHICAL CONSIDERATIONS

The Ethics Committee of UiTM and Medical Research Ethics Committee (MREC) of the Ministry of Health (MOH) approves the study protocol. Permission from the Family Health Development Division (FHDD) of the MOH and the respective Health District Offices are also obtained prior to the conduct of the study. The study is conducted in accordance to the Declaration of Helsinki and Good Clinical Practice (GCP) requirements. Patient information sheet are given and informed consent are obtained from all participants prior to their study enrolment. For participants who are unable to read, the content of the consent form is read aloud to them and a copy of the patient information sheet is given to their next of kin with additional explanation given if needed. Confidentiality of personal information is ensured at all times. Subject enrolment is done by the investigators and not their attending doctors to reduce subject's vulnerability to participate in the study. Subjects are informed of any immediate results obtained from the study that may affect their care or health.

DISCUSSION

The EMPOWER-PAR is the first pragmatic, randomised controlled trial of multifaceted chronic disease management strategies being conducted in the Malaysian public primary care setting. It is expected to yield important new evidence on the improvements of T2DM and HPT clinical outcomes, the two most prevalent chronic diseases being managed in the public primary care sector.

Ultimately, results from this study will provide objective evidence of the effectiveness and cost-effectiveness of a multifaceted intervention based on the CCM in a resource-constrained public primary care setting. If proven effective, the results may be generalisable to other Malaysian public primary clinics which share the same characteristics and would probably be inexpensive to replicate. It is hoped that the objective evidence from EMPOWER-PAR would provide a platform to instigate the much needed primary health care system change in Malaysia.

ELIGIBILITY:
Inclusion criteria

Males and females aged ≥ 18 years who are diagnosed with:

1. T2DM or HPT or both
2. Seen at least once in the last one year at the primary care clinic for the above conditions

Exclusion criteria

1. Type 1 Diabetes Mellitus
2. Receiving renal dialysis
3. Presenting with severe HPT (Systolic BP >180mmHg and/or Diastolic BP >110 mmHg)
4. Diagnosed with conditions resulting in secondary hypertension
5. Diagnosed to have circulatory disorders needing referral to secondary care over the last 1 year e.g. unstable angina, heart attack, stroke, transient ischaemic attacks
6. Receiving shared care between primary and secondary care for complications of T2DM and/or HPT
7. Pregnancy
8. Enrolled in another study

All patients in the intervention arm are required to be seen at least twice by the CDM team of each clinic during the 1-year intervention period. Those who do not comply are considered as lost to follow-up. There is no limit to the number of clinic visits a patient is allowed to make in either arm during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1545 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of patients achieving glycaemic and BP control | 1 year
  Outcome measures are obtained from both intervention and control clinics at baseline and at 1-year after the commencement of intervention.
  Primary Outcomes
  For T2DM patients, primary outcome is measured by the change in the proportion of patients achieving glycaemic target of HbA1c < 6.5%.
  For HPT patients without T2DM, primary outcome is measured by the change in the proportion of patients achieving BP target of < 140/90 mmHg.

SECONDARY OUTCOMES:
Change in the proportion of patients achieving clinical targets: | 1 year
  Change in the proportion of patients achieving target:
  * BP of ≤ 130/80 mmHg (for T2DM patients)
  * Body Mass Index (BMI) < 23 kg/m2
  * Waist Circumference (WC) < 90 cm (men), < 80 cm (women)
  * Total cholesterol [TC] ≤ 4.5 mmol/L
  * Triglycerides [TG] ≤ 1.7 mmol/L
  * Low density lipoprotein [LDL-C] ≤ 2.6 mmol/L
  * High density lipoprotein [HDL-C] ≥ 1.1 mmol/L
Other secondary outcome measures | 1 year
  Other secondary outcome measures include:
  * Change in the Process of Care related to the management of T2DM and HPT
  * Change in the medication adherence level as measured by the 8-item Morisky Medication Adherence Scale (MMAS-8)
  * Change in the prescribing patterns of antihypertensive agents, oral hypoglycaemic agents, insulin usage and lipid lowering agents
  * Patients' perception and experience in receiving care for chronic conditions as measured by the Patients Assessment of Chronic Illness Care (PACIC) score
  * Health care providers' perception, attitude, experience and perceived barriers in implementing the EMPOWER-PAR intervention as measured by qualitative analysis
  * Cost-effectiveness of the EMPOWER-PAR intervention

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Dr. Anis Safura Ramli, MRCGP (UK), Principal Investigator — University Teknologi MARA, Malaysia; Dr. Jamaiyah Haniff, MPH, Principal Investigator — Clinical Research Centre; Dr. Sharmila Lakshmanan, MBBS, Study Director — Clinical Research Centre
Locations (1):
- Universiti Teknologi MARA, Batu Caves, Selangor, Malaysia

REFERENCES:
- [Derived] Ramli AS, Selvarajah S, Daud MH, Haniff J, Abdul-Razak S, Tg-Abu-Bakar-Sidik TM, Bujang MA, Chew BH, Rahman T, Tong SF, Shafie AA, Lee VK, Ng KK, Ariffin F, Abdul-Hamid H, Mazapuspavina MY, Mat-Nasir N, Chan CW, Yong-Rafidah AR, Ismail M, Lakshmanan S, Low WH; EMPOWER-PAR Investigators. Effectiveness of the EMPOWER-PAR Intervention in Improving Clinical Outcomes of Type 2 Diabetes Mellitus in Primary Care: A Pragmatic Cluster Randomised Controlled Trial. BMC Fam Pract. 2016 Nov 14;17(1):157. doi: 10.1186/s12875-016-0557-1. PMID 27842495
- [Derived] Ramli AS, Lakshmanan S, Haniff J, Selvarajah S, Tong SF, Bujang MA, Abdul-Razak S, Shafie AA, Lee VK, Abdul-Rahman TH, Daud MH, Ng KK, Ariffin F, Abdul-Hamid H, Mazapuspavina MY, Mat-Nasir N, Miskan M, Stanley-Ponniah JP, Ismail M, Chan CW, Abdul-Rahman YR, Chew BH, Low WH. Study protocol of EMPOWER participatory action research (EMPOWER-PAR): a pragmatic cluster randomised controlled trial of multifaceted chronic disease management strategies to improve diabetes and hypertension outcomes in primary care. BMC Fam Pract. 2014 Sep 13;15:151. doi: 10.1186/1471-2296-15-151. PMID 25218689